CLINICAL TRIAL: NCT01873638
Title: Comparing Minilaparotomy and Laparoscopic Cholecystectomy as a Day Surgery Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Matti Eskelinen, professor, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KUH5200630
Record Dates: First submitted 2013-06-04; First posted 2013-06-10 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-06

CONDITIONS: Gallstone Disease
Keywords: 5-year outcome after cholecystectomy
MeSH Terms: conditions — Cholelithiasis | interventions — Cholecystectomy

ARMS (2):
- Minilaparotomy (Other): Minilaparotomy cholecystectomy as a day surgery
  Interventions: Procedure: Cholecystectomy
- Laparoscopy (Other): Laparoscopic cholecystectomy as a day surgery
  Interventions: Procedure: Cholecystectomy

INTERVENTIONS:
Procedure: Cholecystectomy

SUMMARY:
Minlaparotomy (MC) and laparoscopic cholecystoctomy (LC) are commonly applied surgical techniques for the management of symptomatic gallstone disease and both techiques have shown to be feasible for day surgery. However, to our knowledge the long-term outcome between these approaches has not been compared in randomised trials as day surgery procedures.

ELIGIBILITY:
Inclusion Criteria:

* Cholelithiasis confirmed by preoperative ulrasound
* No significant co-morbidities
* The ASA physical status classification 1 or 2
* Age 18 to 65 yrs.
* BMI less than 35
* Less than a one hour journey from hospital to home
* Patient´s own motivation to daysurgery

Exclusion Criteria:

* Elevated liver laboratory tests
* Earlier jaundice
* A suspicion or verified stones in the common bile duct
* Acute cholecystitis
* A history of pancreatitis
* Hepatic cirrhosis
* Suspicion of cancer
* Previous open upper abdominal surgery
* Asthma
* Peptic ulcer
* Bleeding disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-02; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Chronic post-surgical pain | Five year outcome

SECONDARY OUTCOMES:
Quality of life | Five year outcome

OTHER OUTCOMES:
Cosmetic satisfaction | Five year outcome
Residual abdominal symptoms | Five year outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Kuopio University Hospital, Kuopio, Northern Savonia, Finland